CLINICAL TRIAL: NCT05921812
Title: Biochemical Role of Circulating microRNAs Expression as Diagnostic Markers for Non-Hodgkin's Lymphoma Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shrouk Mostafa Galal, demonstrator at medical biochemistry department, Sohag University
Other Study IDs: Soh-Med-23-06-03MS
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: apparently healthy individuals with no chronic illness
  Interventions: Diagnostic Test: real time pcr
- cases: newly diagnosed Non-Hodgkin's lymphoma patients
  Interventions: Diagnostic Test: real time pcr

INTERVENTIONS:
Diagnostic Test: real time pcr — evaluate the expression of certain circulating microRNAs by real time pcr

SUMMARY:
Lymphomas are a fairly common malignancy accounting for approximately half of all newly diagnosed hematological neoplasms, and they comprise the sixth most common group of malignancies worldwide in both men and women, With marked geographic variations and affecting more males than females within the age range of 1 to 85 years but peaking within the second decades of life (Oluwasola AO et al., 2011, Roman E et al., 2011 and Jemal A et al., 2010) . Lymphomas have traditionally been classified as either Hodgkin's lymphoma (HL) or non-Hodgkin's lymphoma (NHL) based on the presence or absence of the Reed-Sternberg (RS) cell on histology. (Fitzmaurice C et al., 2017). Non-Hodgkin's lymphoma (NHLs) comprise a wide class of lymphoid neoplasms that evolve from the clonal expansion of mature B, T and natural killer (NK) cells in different stages of development (Morton, L.M. et al., 2014 and Schmitz R et al., 2009). NHLs are the most prevalent hematopoietic neoplasms, accounting for approximately 4.3% of all cancer diagnoses (Sant, M. et al., 2010) , Of them, B cell NHL accounts for approximately 30% of all lymphoid neoplasms, followed by HL (8%) and T/NK neoplasms (5%) (Morton, L.M. et al., 2006).

MicroRNAs (miRNAs) are a class of small, naturally occurring, noncoding and single-stranded RNA molecules (18, 22 nucleotides) that function as post-transcriptional regulators by directly cleaving target messenger RNA (mRNA) or translational repression (Bartel DP. Et al., 2004). The discovery of miRNA has exposed a new layer of gene expression regulation that affects many physiological and pathological processes of life (Lawrie CH. Et al., 2013).

Many abnormal miRNA expression patterns are found in various human malignancies, and certain miRNAs play roles as oncogenes or tumor suppressors (Ling N et al., 2013). Certain miRNAs have been found to characterize various subtypes of NHL and have important roles in B-cell differentiation and lymphomagenesis (Zhang J et al., 2009, Malumbres R et al., 2009, Basso K et al., 2009 and Auer RL et al., 2011). Recently, many studies had shown that tumor cell-specific miRNAs were detectable in the plasma and serum of patients with cancer. Therefore, miRNAs may be served as good biomarkers for early detection, diagnosis, and follow up of patients with cancer (Cortez MA et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

1. This study will include patients who have newly diagnosed, histo-pathologically proved Non-Hodgkin's lymphoma.
2. Age from 18 to 75 years old.
3. anti-neoplastic treatment naïve patients.
4. No associated other malignancies (neither Synchronous nor metachronous) than Non-Hodgkin's lymphoma.

Exclusion Criteria:

1. children below 18 years old or elderly people more than 75 years old
2. patients not newly diagnosed with non-Hodgkin's lymphoma
3. presence of any associated other malignancies than non-Hodgkin's lymphoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have newly diagnosed, histo-pathologically proved Non-Hodgkin's lymphoma,aged from 18-75 and healthy control of matched age and sex
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
microRNA16-1 | 6 months
  quantification of microRNA16-1 by real time PCR in Non-Hodgkin's lymphoma patients
microRNA 21 | 6months
  quantification of microRNA 21 by real time PCR in Non-Hodgkin's lymphoma patients
microRNA 155 | 6 months
  quantification of microRNA155 by real time PCR in Non-Hodgkin's lymphoma patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

REFERENCES:
- [Background] Sun CM, Luan CF. Overexpression of microRNA-21 in peripheral blood mononuclear cells of patients with B-cell non-Hodgkin's lymphoma is associated with disease stage and treatment outcome. Eur Rev Med Pharmacol Sci. 2015 Sep;19(18):3397-402. PMID 26439034
- [Background] Jorgensen S, Paulsen IW, Hansen JW, Tholstrup D, Hother C, Sorensen E, Petersen MS, Nielsen KR, Rostgaard K, Larsen MAH, Brown PN, Ralfkiaer E, Homburg KM, Hjalgrim H, Erikstrup C, Ullum H, Troelsen J, Gronbaek K, Pedersen OB. The value of circulating microRNAs for early diagnosis of B-cell lymphoma: A case-control study on historical samples. Sci Rep. 2020 Jun 15;10(1):9637. doi: 10.1038/s41598-020-66062-1. PMID 32541886
- [Background] Bedewy AML, Elmaghraby SM, Shehata AA, Kandil NS. Prognostic Value of miRNA-155 Expression in B-Cell Non-Hodgkin Lymphoma. Turk J Haematol. 2017 Aug 2;34(3):207-212. doi: 10.4274/tjh.2016.0286. Epub 2017 Feb 1. PMID 28148469
- [Background] Fang C, Zhu DX, Dong HJ, Zhou ZJ, Wang YH, Liu L, Fan L, Miao KR, Liu P, Xu W, Li JY. Serum microRNAs are promising novel biomarkers for diffuse large B cell lymphoma. Ann Hematol. 2012 Apr;91(4):553-9. doi: 10.1007/s00277-011-1350-9. Epub 2011 Oct 11. PMID 21987025